CLINICAL TRIAL: NCT05171491
Title: Clinical Evaluation of LungLB in Subjects Presenting With Indeterminate Pulmonary Nodules
Brief Title: LungLB in Subjects Presenting With Indeterminate Pulmonary Nodules
Status: Active, not recruiting | Type: Observational
Sponsor: LungLife AI (Industry)
Responsible Party: Sponsor
Other Study IDs: LAI-001
Record Dates: First submitted 2021-11-12; First posted 2021-12-29 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodules
Keywords: Lung Cancer; Circulating Genetically Abnormal Cells (CGAC); 4-color FISH; Increased/Decreased Risk; Early Lung Cancer Detection; Indeterminate Nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White blood cells and plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indeterminate Lung Nodule: Subjects that present with indeterminate lung nodules at time of biopsy. No intervention outside of standard of care.

SUMMARY:
Correlate performance of LungLB Test with outcome of a scheduled biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old with a CT identified indeterminate pulmonary nodule and scheduled for biopsy, at the time of consent.
2. Planned biopsy nodule of interest:

   1. is solid ≤3 cm; or
   2. is nonsolid, ground glass opacity, of any size; or
   3. is part solid, where the solid component is no larger than 3cm (maximum diameter).

Exclusion Criteria:

1. Current and or prior diagnosis +/- treatment of non-lung cancer within the past 3 years.
2. Current and or prior lung cancer diagnosis within 2 years following intent-to-cure surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with suspicious indeterminate pulmonary nodules identified incidentally or through a lung cancer screening program. up to 15 institutions geographically distributed across the US.
Sampling Method: Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of LungLB test as compared to results from a tissue/FNA biopsy. | up to 60 days

SECONDARY OUTCOMES:
Evaluate Clinical Variables With and Without LungLB Test Results | up to 60 days
  Evaluate the independent and associated contribution of readily available clinical variables including age, race, gender, socioeconomic level, environmental exposure, tobacco use, and radiology data combined with and without the LungLB test results and correlate with biopsy (tissue / FNA) outcome of indeterminate pulmonary nodules.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donovan, MD, Study Director — LungLife AI
Locations (12):
- United States (12):
  - Clinical Site 04, Los Angeles, California
  - Clinical Site 05, Bay Pines, Florida
  - Clinical Site 03, Miami, Florida
  - Clinical Site 07, Hines, Illinois
  - Clinical Site 27, Kansas City, Kansas
  - Clinical Site 12, Wichita, Kansas
  - Clinical Site 08, Kansas City, Missouri
  - Clinical Site 18, Reno, Nevada
  - Clinical Site 01, New York, New York
  - Clinical Site 25, Columbia, South Carolina
  - Clinical Site 02, Houston, Texas
  - Clinical Site 32, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No